CLINICAL TRIAL: NCT03957395
Title: Comparison of Effectiveness of Tonic, High Frequency and Burst Spinal Cord Stimulation in Chronic Pain Syndromes: a Double-blind, Randomised, Cross-over, Placebo Controlled Trial
Brief Title: Comparison of Effectiveness of Tonic, High Frequency and Burst Spinal Cord Stimulation in Chronic Pain Syndromes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jan Biziel University Hospital No 2 in Bydgoszcz (Other)
Responsible Party: Principal Investigator, Pawel Sokal, Head of Department of Neurosurgery and Neurology, Jan Biziel University Hospital No 2 in Bydgoszcz
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: JBUH-NN-SCS-2018
Record Dates: First submitted 2019-05-17; First posted 2019-05-21 (Actual); Last update posted 2019-05-29 (Actual); Status verified 2019-05

CONDITIONS: Failed Back Surgery Syndrome; CRPS (Complex Regional Pain Syndromes)
Keywords: FBSS; CRPS; SCS; Burst; Tonic; High-frequency
MeSH Terms: conditions — Failed Back Surgery Syndrome; Complex Regional Pain Syndromes

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- scs high-frequency (Experimental): high-frequency stimulation
  Interventions: Device: Device: Precision Novi™ system Neurostimulation procedures
- scs tonic (Experimental): tonic stimulation
  Interventions: Device: Device: Precision Novi™ system Neurostimulation procedures
- scs burst (Experimental): burst stimulation
  Interventions: Device: Device: Precision Novi™ system Neurostimulation procedures
- scs off (Placebo Comparator): off stimulation
  Interventions: Device: Device: Precision Novi™ system Neurostimulation procedures

INTERVENTIONS:
Device: Device: Precision Novi™ system Neurostimulation procedures — SCS with Device: Precision Novi™ system
  Other Names: SCS

SUMMARY:
Spinal cord stimulation (SCS) is one of the most commonly undertaken neuromodulatory surgery techniques in the treatment of neuropathic pain. The indication for SCS is an ineffective conservative treatment of chronic pain syndromes. The effectiveness of SCS in the case of neuropathic pain is high. The positive result of SCS treatment is the reduction of previous painful symptoms by min. 50% and / or a reduction in the amount of taken analgesics and an improvement in the quality of life including sleep quality. Long-term studies estimate that in a properly selected group of patients more than 50% of patients achieve pain reduction by the required 50% and about 60% - 70% have an improvement in the quality of life and a reduction of pain.

The efficacy of SCS in different modes of stimulation is evaluated. Patients receive four different types of stimulation for 2-week period - not knowing what kind of stimulation it is. It is said that in one type of stimulation they would feel parestesias and in other three they would not. Patients are not informed that beside tonic, burst and high frequency stimulation, the fourth is an off stimulation to check for placebo effect. The test is double-blinded

DETAILED DESCRIPTION:
Patients with FBSS and CRPS are evaluated for VAS,, dissability scale, Quality of Life (QoL), sleep disorders and mental disorders.

All patients undergo percutaneus (1 or 2) 8-contact SCS electrode implantation with trial.

All patients are blindly randomized to tonic or burst or high frequency or off stimulation. After 2-week period each participant is adequately switched to another type of stimulation for next 2 weeks. Alltogether crossover takes 8 weeks: four 2-week periods of tonic, burst, HF and off stimulation. At the end of trial period patients are subjected to the mode of stimulation which is the most efficent. The final 2-week stimulation is performed with final renewed evaluation for VAS, amount of taken medications, dissability scale, Quality of Life (QoL), sleep disorders and mental disorders. Follow-up observation will last up to 12 months.

ELIGIBILITY:
Inclusion Criteria:

1. FBSS, CRPS patients with neuropathic and mixed pain in low-back and/or legs refractory to conservative therapy
2. Chronic pain as a result of FBSS that exists for at least 6 months
3. ≥ 18 years of age
4. Written consent of the patient to participate in study procedures.

Exclusion Criteria:

1. Active malignancy
2. Addiction to any of the following: drugs, alcohol and/or medication
3. Evidence of an active disruptive psychiatric disorder or other known condition significant enough to impact perception of pain, compliance to intervention and/or ability to evaluate treatment outcome as determined by investigator
4. Local infection or other skin disorder at site of surgical incision
5. Pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2018-09-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Scale | 12 months
  Change from baseline in VAS for back and leg pain
Oswestry Disability Index | 12 months
  Change from baseline in functionality using the ODI score
Adverse Events | 12 months
  Number of AE through the study
Number of pain medication | 12months
  List of pain medication taken by patient
Quality of life scale | 12months
  Quality of life assessed by EuroQol group - 5 Dimensions (EQ-5D)

CONTACTS AND LOCATIONS:
Overall Officials: Paweł Sokal, Principal Investigator — Jan Biziel University Hospital
Locations (1):
- Department of Neurosurgery and Neurology University Hospital nr 2 Collegium Medicum Nicolaus Copernicus University, Bydgoszcz, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] O'Connell NE, Ferraro MC, Gibson W, Rice AS, Vase L, Coyle D, Eccleston C. Implanted spinal neuromodulation interventions for chronic pain in adults. Cochrane Database Syst Rev. 2021 Dec 2;12(12):CD013756. doi: 10.1002/14651858.CD013756.pub2. PMID 34854473